CLINICAL TRIAL: NCT02709629
Title: The Effects of Computerized Cognitive Training on Diabetic Elderly, Who Are at High Risk for Dementia
Brief Title: CCT for Older Diabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Dr. Alex Bahar-Fuchs, Dr Alex Bahar-Fuchs, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0573-13-SMC
Record Dates: First submitted 2016-02-25; First posted 2016-03-16 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Older Diabetic Persons Without Dementia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized and adaptive computerised cognitive training (Experimental): Training in this group is individualized using a computer algorithm which assigns tasks (from a pool of 33 training tasks) on the basis of cognitive strengths and weaknesses as determined by the training program. In addition, task difficulty is adaptive and responsive to performance level. Participants are able to see feedback on their progress each training session in the form of a session-score. A range of behavior change techniques are used throughout the training period (delivered via scheduled monitoring phone calls, and email contact with participants) to support the compliance and adherence of participants. These include a range of motivation and confidence building strategies, based on a theoretical framework. Participants are required to train for approx. 30 min., 3 times per week, for 8 weeks.
  Interventions: Behavioral: Individualized and adaptive computerized cognitive training
- Active control (Active Comparator): Training in this group is generic, and tasks (from the same pool of 33 training tasks) are randomly selected by the training program. In addition, task difficulty is fixed, such that irrespective of performance, each time a participant is presented with a given task, the level of difficulty returns to the basic level. Participants in this arm do not receive feedback on their progress at the end of each training session. The same protocol of behavior change techniques is used in this intervention arm.
  Participants are also required to train for approx. 30 min., 3 times per week, for 8 weeks.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Individualized and adaptive computerized cognitive training
  Arms: Individualized and adaptive computerised cognitive training
Behavioral: Active control
  Arms: Active control

SUMMARY:
The current study examines the efficiency of a home-based computerized cognitive training (CT) intervention targeting older adults with diabetes.The primary aim of the study is to evaluate the effects of CCT on cognitive and disease management in non-demented older diabetes adults. Investigators will also evaluate the effect of the intervention on a range of secondary outcomes, including mood, caregiver burden, self-efficacy, and for a small sub-sample, on brain activity as reflected in changes in task-related blood-flow on fMRI.

DETAILED DESCRIPTION:
Evidence suggests a link between diabetes-related processes and increased risk of cognitive decline and dementia in older adults. Optimal disease self-management may be key in the prevention of cognitive decline among older diabetic patients, but this may be compromised due to sub-clinical cognitive impairment.

In the current study, 120 community-dwelling, non-demented participants aged 65 and over, with a diagnosis of Type 2 diabetes will be randomly assigned either to an 8-week, home-based individually-tailored CCT program with adaptive difficulty level, and regular performance feedback, or to an 8-week, home-based active control (AC) condition, involving training on a generic CCT program with fixed difficulty level and without performance feedback. Both intervention groups also include a range of theory-informed behavior change techniques (BCTs), including self-efficacy management, self-monitoring and goal-setting in order to enhance treatment fidelity, and to maximize treatment compliance and adherence. In both groups, participants train approx. 30 min. per day, 3 times per-week for 8-weeks. Participants undergo a comprehensive evaluation of all outcomes at baseline, immediately after the intervention, and at a 6-month follow-up, with 1-week booster training completed 3 months from completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over
* diagnosis of type 2 diabetes
* Health cover provided by Maccabi Health Services (MHS)
* Access to a home computer and internet connection
* Availability of a close relative/informant with regular and frequent contact with the participant (at least 10 hours per week), willing to respond to questionnaires at all time points.
* Fluency in Hebrew or English
* Living in the Tel-Aviv metropolitan area and surrounds

Exclusion Criteria:

* An existing diagnosis of dementia
* Prescription of dementia-related medication.
* Participation in a previous cognitive intervention study in the preceding year.
* Significant hearing/vision impairment likely to interfere with assessment and/or training
* Significant psychiatric/neurological or medical issues that may affect cognitive function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in global cognition as reflected in a composite cognitive score at 9 weeks | 9 weeks
Change from baseline in diabetes self management as reflected in the diabetes self-management questionnaire | 9 weeks

SECONDARY OUTCOMES:
Change in domain-specific cognitive abilities (memory, non-memory) measured by composite scores from the neuropsychological test battery, at 9 weeks | 9 weeks(immediately post-intervention)
Change in domain-specific cognitive abilities (memory, non-memory) measured by composite scores from the neuropsychological test battery, at 35 weeks | 35 weeks (6 months follow up)
Change in meta-memory (subjective ratings of memory performance) as reflect on the Meta-Memory Questionnaire at 9 weeks | 9 weeks
Change in meta-memory (subjective ratings of memory performance), as reflect on the Meta-Memory Questionnaire, at 35 weeks | 35 weeks (6 months follow up)
Change in self-reported mood-related symptoms on the geriatric depression scale at 9 weeks | 9 weeks
Change in self-reported mood-related symptoms on the geriatric depression scale at 35 weeks | 35 weeks (6 months follow up)
Change in informant-reported care-giving burden on the Zarit Burden Interview at 9 weeks | 9 weeks
Change in informant-reported care-giving burden on the Zarit Burden Interview at 35 weeks | 35 weeks (6 months follow up)
Change in blood sugar levels on a blood glucose test at 35 weeks | 35 weeks
Change from baseline in global cognition as reflected in a composite cognitive score at 35 weeks | 35 weeks
Change from baseline in diabetes self-management as reflected in scores on the diabetes self-management questionnaire at 35 weeks | 35 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Joseph Sagol Neuroscience Center, Sheba Medical Center, Ramat Gan, Australian National University, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bahar-Fuchs A, Barendse MEA, Bloom R, Ravona-Springer R, Heymann A, Dabush H, Bar L, Slater-Barkan S, Rassovsky Y, Schnaider Beeri M. Computerized Cognitive Training for Older Adults at Higher Dementia Risk due to Diabetes: Findings From a Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2020 Mar 9;75(4):747-754. doi: 10.1093/gerona/glz073. PMID 30868154